CLINICAL TRIAL: NCT04108091
Title: Vyndaqel Capsules Special Investigation - Investigation on Patients With Transthyretin Amyloid Cardiomyopathy
Brief Title: Vyndaqel Capsules Special Investigation (ATTR-CM)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461064; NCT04108091 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Transthyretin (TTR) Amyloid Cardiomyopathy
Keywords: transthyretin amyloid cardiomyopathy;; TTR Cardiomyopathy;; Transthyretin (TTR) Amyloid Cardiomyopathy;; Vyndaqel;; Tafamidis meglumine;; ATTR-CM;; Vynmac;
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Therapeutics; tafamidis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment for TTR amyloidosis: Transthyretin amyloid cardiomyopathy (wild-type or variants) patients administered Vyndaqel and Vynmac.
  Interventions: Drug: Treatment for TTR amyloidosis

INTERVENTIONS:
Drug: Treatment for TTR amyloidosis — The usual adult dose is 80 mg of Tafamidis Meglumine orally once daily. The dose may be reduced if not tolerated.
  Other Names: Vyndaqel
Drug: Treatment for TTR amyloidosis — The usual adult dose is 61 mg of tafamidis orally once daily.
  Other Names: Vynmac

SUMMARY:
Secondary Data Collection : To confirm the safety and effectiveness profiles under the actual medical practice of Vyndaqel in Japan. This study is conducted in accordance with the protocol even when Vynmac is used, and information the use of Vynmac during the observation period is also collected.

DETAILED DESCRIPTION:
To comprehend information on the long-term safety (e.g., onset status of adverse reactions), etc. of patients who are treated with Vyndaqel for the treatment of transthyretin amyloid cardiomyopathy. When Vynmac is used, conduct the study to grasp information on safety (e.g., onset status of adverse reactions),etc. during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Patients administered Vyndaqel for the treatment of ATTR-CM

Exclusion Criteria:

* N/A

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are administered with this drug for the treatment of ATTR-CM
Sampling Method: Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse drug reaction | 30 months

SECONDARY OUTCOMES:
Number of survival | 30months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461064